CLINICAL TRIAL: NCT00043121
Title: A Phase I Study of Oxaliplatin, 5-Fluorouracil, and Leucovorin in Combination With Oral Capecitabine in Patients With Advanced Malignancy
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Cancer That is Metastatic or Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00004; NCI-2013-00004 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-5904; WCCC-CO-02901; CO 02901 (Other: University of Wisconsin Hospital and Clinics); 5904 (Other: CTEP); U01CA062491 (NIH)
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Oxaliplatin; Leucovorin; Fluorouracil; Capecitabine

ARMS (1):
- Treatment (combination chemotherapy) (Experimental): Patients receive oxaliplatin IV over 2 hours, leucovorin calcium IV, and fluorouracil IV on days 1 and 15. Patients also receive oral capecitabine every 8 hours on days 1-2 and 15-16. Leucovorin calcium and fluorouracil administration is held at dose level 4 and above. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: oxaliplatin; Drug: leucovorin calcium; Drug: fluorouracil; Drug: capecitabine; Other: pharmacological study

INTERVENTIONS:
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Drug: capecitabine — Given orally
  Other Names: CAPE; Ro 09-1978/000; Xeloda
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial studies the side effects and best dose of capecitabine when given together with oxaliplatin, leucovorin calcium, and fluorouracil in treating patients with advanced cancer that is metastatic or cannot be removed by surgery. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the MTD and toxicity profile of oral capecitabine in combination with q 2 weekly intravenous oxaliplatin in patients with advanced malignancies.

SECONDARY OBJECTIVES:

I. To characterize the pharmacokinetic parameters of capecitabine at the recommended phase II dose for combinations of capecitabine, oxaliplatin, 5-fluorouracil, and leucovorin, as well as for the combination of capecitabine and oxaliplatin.

II. To observe for and record any antitumor activity.

OUTLINE: This is a dose-escalation study of capecitabine.

Patients receive oxaliplatin IV over 2 hours, leucovorin calcium IV, and fluorouracil IV on days 1 and 15. Patients also receive oral capecitabine every 8 hours on days 1-2 and 15-16. Leucovorin calcium and fluorouracil administration is held at dose level 4 and above. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed malignancy which is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* There is no limit on prior therapies
* ECOG performance status 0-2
* Leukocytes >= 3,000/ul
* Absolute neutrophil count >= 1,500/ul
* Platelets >= 100,000/ul
* Total bilirubin =< 1.5 mg/dL
* AST (SGOT)/ALT (SGPT) =< 2.5 x institutional upper limit of normal
* Creatinine clearance >= 50 mL/min as calculated by the Cockroft-Gault formula
* Patients with no >= grade 2 (Common Toxicity Criteria [CTC] 2.0) neuropathy
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Breastfeeding should be discontinued if the mother is treated with oxaliplatin
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study
* Patients undergoing therapy with other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other toxicities
* History of allergy to platinum compounds or to antiemetics appropriate for administration in conjunction with protocol-directed chemotherapy
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, or unstable angina pectoris, or cardiac arrhythmia
* Pregnant and nursing women are excluded from this study because oxaliplatin is a DNA alkylating agent with the potential for teratogenic or abortifacient effects
* Human immunodeficiency virus (HIV)-positive patients receiving anti-retroviral therapy (HAART) are excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2002-06; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
MTD, defined as the highest dose level which results in DLT in fewer than 2/6 patients, graded according to the NCI CTC version 2.0 | Up to 28 days

SECONDARY OUTCOMES:
Incidence of adverse events, graded according to NCI CTC version 2.0 | Up to 6 years
Overall survival | Up to 6 years
  Estimated using the product-limit method of Kaplan and Meier.
Time to progression | Up to 6 years
  Estimated using the product-limit method of Kaplan and Meier.
Duration of response | Up to 6 years
  Estimated using the product-limit method of Kaplan and Meier.

CONTACTS AND LOCATIONS:
Overall Officials: George Wilding, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States